CLINICAL TRIAL: NCT03099889
Title: Women's Health Initiative Strong and Healthy Exercise Trial-2-Prevent Heart Failure
Brief Title: WHISH-2-Prevent Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Stanford University (Other); Ohio State University (Other); Fred Hutchinson Cancer Center (Other); University of North Carolina, Chapel Hill (Other); University of California, San Francisco (Other); University of California, San Diego (Other); University at Buffalo (Other); Wake Forest University (Other)
Responsible Party: Principal Investigator, Charles B. Eaton, Principal Investigator, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5R01HL130591-02 (NIH)
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Physical Activity; Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Normal Ejection Fraction; Strength Training; Elderly; Women
MeSH Terms: conditions — Motor Activity; Heart Failure | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized consent design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant in intervention arm signed an informed consent umasking the exercise intervention, participants in the control arm have already consented to ongoing outcomes assessment and yearly surveys regarding physical activity and other lifestyle activities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity intervention arm (Experimental): Receive a tailored behavioral interventions for exercise and strength training via multiple channels including frequent mailings, integrated voice response and outreach phone calls, interactive website, and referral to local community exercise resources.
  Interventions: Behavioral: Physical Activity
- Control arm (No Intervention): Receive general health mailings

INTERVENTIONS:
Behavioral: Physical Activity — Physical activity intervention based upon stage of change and social cognitive theory based interventions
  Arms: Physical Activity intervention arm

SUMMARY:
The WHISH-2-Prevent Heart Failure (HF) study is an ancillary study to the Women's Health Initiative Strong and Healthy (WHISH) exercise pragmatic trial. The WHISH-2-Prevent HF trial examines the intervention effect of physical activity (PA) on both incident HF and HF burden (recurrent HF and CVD death in those with HF) in a cost effective manner in elderly women. In addition, it will allow a dose-finding analysis to better understand the type, intensity and frequency of PA that leads to a reduced risk and burden of HF. The focus of the parent WHISH trial is on atherosclerotic cardiovascular disease and not heart failure.

DETAILED DESCRIPTION:
A recently funded large pragmatic PA trial, Women's Health Initiative Strong and Healthy (WHISH) trial based upon two decades of PA intervention experience using enhanced communication and behavioral techniques, has randomized 49,936 elderly women (average age 79) and will evaluate its intervention effect on the risk of atherosclerotic CVD. This translational intervention is aimed at reducing sedentary time and achieving or maintaining aerobic and strength enhancing PA levels currently recommended for cardiovascular benefit. The WHISH-2-Prevent HF, represents the first and largest primary prevention exercise trial ever performed focusing on HF and will examine the intervention effect of PA , on both incident HF and HF burden (recurrent HF and CVD death in those with HF) in a cost effective manner in elderly women. In addition, it will allow a dose-finding analysis to better understand the type, intensity and frequency of PA that leads to a reduced risk and burden of HF.

Aim 1: Test whether older women who are initially free of HF and randomized to a translational PA intervention will reduce the rate of incident HF compared to those not randomized to the translational PA intervention.

H1: Women free of HF randomized to the PA intervention will have reduced rates of incident HF compared to those not randomized.

Aim 2: Test whether older women with and without HF at baseline randomized to a translational PA intervention will reduce the HF burden (number of acute HF hospitalizations and CVD death in those with antecedent HF) compared to those not randomized to the translational PA intervention. H2: Women randomized to the PA intervention will have reduced HF Burden compared to those not randomized

Exploratory Aim 3: Analyze the type, intensity and frequency of physical activity including skeletal muscle strengthening associated with a reduced risk of HF and HF burden in elderly women. H3: Women who have low levels of sedentary behavior by either increasing or maintaining light intensity or moderate intensity physical activity will have reduced rates of HF compared to women who remain sedentary. Those that add skeletal muscle strengthening will have additional benefits.

ELIGIBILITY:
Inclusion Criteria:

* alive, community dwelling,

Exclusion Criteria:

* Dementia, need walking aide, reside in nursing home

Ages: 66 Years to 102 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — self-identified as post-menopausal women and participate in the women's health initiative study
Enrollment: 49936 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
hospitalized heart failure | within 4 years of randomization
  first acute decompensated hospitalized heart failure event

SECONDARY OUTCOMES:
Heart failure with reduced ejection fraction | within 4 years of randomization
  reduced systolic function on echo or other objective imaging
Heart failure with preserved ejection fraction | within 4 years of randomization
  normal systolic function on echo or other objective imaging
Recurrent hospitalized heart failure | within 4 years of randomization
  number of acute decompensated heart failure events
Cardiovascular disease mortality | within 4 years of randomization
  Underlying cause of death was either heart failure or cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Eaton, MD, MS, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Within two years of completion of study, de-identified data will be made available via WHI website after approval by the Publications and Presentation committee and data use agreement signed